CLINICAL TRIAL: NCT06071169
Title: The Effect of Progressive Relaxation Exercise on Nurses' Life Satisfaction, Comfort and Burnout Levels
Brief Title: The Effect of Progressive Relaxation Exercise on Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Instructor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 47/2023
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Progressive Relaxation Exercise; Comfort; Life Satisfaction; Burnout
MeSH Terms: conditions — Personal Satisfaction; Burnout, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): progressive relaxation exercise group The nurses will perform the relaxation exercises 3 days a week for 5 weeks, 20 minutes in each practice.
  Interventions: Other: progressive relaxation exercise
- Control (No Intervention): Control group No application has been made.

INTERVENTIONS:
Other: progressive relaxation exercise — Nurses will be asked to perform relaxation exercises 3 days a week for 5 weeks, 20 minutes in each practice.
  Arms: Intervention

SUMMARY:
This study aims to examine the effect of progressive relaxation exercise on nurses' life satisfaction, comfort and burnout levels. Data will be collected by using Descriptive Characteristics Information Form, Satisfaction with Life Scale, Nurse Comfort Scale and Burnout Scale. The nurses in the intervention group will be asked to perform relaxation exercises. The nurses in the control group will not receive any intervention.

DETAILED DESCRIPTION:
This study aims to examine the effect of progressive relaxation exercise on nurses' life satisfaction, comfort and burnout levels. This study will be conducted as a randomized controlled experimental study. Data will be collected by using Descriptive Characteristics Information Form, Satisfaction with Life Scale, Nurse Comfort Scale and Burnout Scale. The nurses in the intervention group will be asked to perform relaxation exercises 3 days a week for 5 weeks, 20 minutes in each practice. The nurses in the control group will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

Working as a nurse in a tertiary treatment center for at least 3 years Have not participated in any relaxation exercise Absence of neurological/psychiatric disorders Not having an obstacle to exercise Nurses who volunteered to participate in the study will be included in the study.

Exclusion Criteria:

Individuals who have any exercise program and use any relaxation method (yoga, acupuncture, massage, music therapy, etc.) will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2023-11-27 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Comfort | 5 weeks after first meeting
  The scale consists of 39 items in total. Each statement in the scale has a Likert-type rating ranging from 1-4 from "strongly disagree" to "strongly agree". 24 of the expressions are positive and 15 are negative, and negative items are reversed in scoring. Accordingly, a high score (4) indicates high comfort, a low score (1) indicates low comfort, and a low score (1) indicates high comfort in negative statements, and a high score (4) indicates low comfort. The Cronbach alpha coefficient was found to be 0.915.
Satisfaction with Life | 5 weeks after first meeting
  It was developed to determine an individual's satisfaction with his/her life. The scale consists of five Likert-style items on a 7-point scale (1: strongly disagree, 7: strongly agree). The lowest score that can be obtained from the scale is 5 and the highest score is 35. A low score is accepted as an indicator of low life satisfaction and a high score as an indicator of high life satisfaction.
Burnout | 5 weeks after first meeting
  It was created to measure the perceived burnout level. The scale consists of 22 items in total and is 7-point Likert type. These options are as follows in terms of severity; 1- Never, 2- Very Rarely, 3- Sometimes, 4- Most of the Time, 5- Always. There are three subscales: emotional exhaustion, depersonalization and low personal accomplishment.

IPD SHARING:
Plan to Share IPD: No